CLINICAL TRIAL: NCT00724035
Title: Onset Time of Brachial Plexus Anesthesia With the Axillary or Infraclavicular Approach Under Real-Time Ultrasound Guidance: a Randomized Controlled Trial
Brief Title: Ultrasound-Guided Axillary or Infraclavicular Nerve Block for Upper Limb Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Parma (Other)
Responsible Party: Guido Fanelli, MD, University of Parma
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANEST-ORT-02
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Upper Extremity; Orthopedic Surgery; Trauma; Forearm Injuries; Nerve Block
Keywords: Anesthesia; Upper extremity; Nerve block; Ultrasound; Brachial plexus
MeSH Terms: conditions — Wounds and Injuries; Forearm Injuries | interventions — Midazolam; Benzodiazepines; Premedication; Ropivacaine; Anesthetics, Local; Fentanyl; Analgesics, Opioid; Analgesics; Anesthesia, General; Anesthesia, Conduction; High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infraclavicular (Experimental): This group will receive an ultrasound-guided infraclavicular brachial plexus block.
  Interventions: Drug: Midazolam; Drug: Ropivacaine; Drug: Fentanyl; Procedure: General anesthesia; Procedure: Infraclavicular brachial plexus block
- Axillary (Active Comparator): This group will receive an ultrasound-guided axillary brachial plexus block.
  Interventions: Drug: Midazolam; Drug: Ropivacaine; Drug: Fentanyl; Procedure: General anesthesia; Procedure: Axillary brachial plexus nerve block

INTERVENTIONS:
Drug: Midazolam — Procedural sedation before the execution of the block.
  * 0.03 mg/kg iv bolus
  Other Names: Versed; Benzodiazepine; Premedication; Sedation
Drug: Ropivacaine — 0.75% (wt/vol) solution, 20 ml perineural injection
  Other Names: Naropin; Local anesthetic; Amide local anesthetic
Drug: Fentanyl — 50 µg iv bolus prn for pain during surgery, up to 150 µg
  Other Names: Opioid; Analgesic
Procedure: General anesthesia — General anesthesia will be induced if pain during surgery develops which is intractable with iv fentanyl ≤150 µg.
  Other Names: Monitored anesthesia care
Procedure: Axillary brachial plexus nerve block — Blocks will be performed under high-resolution real-time ultrasound guidance.
  Patients will be in the supine position. With the abducted arm flexed 90° at the elbow, the transducer will scan for the axillary artery in its short-axis. Individual nerves will be sought for around the artery.
  A 22G, 17°-bevel needle will be advanced in-plane to inject aliquots of local anesthetic around each nerve structure up to the prescribed dose.
  Other Names: Peripheral Nerve Block; Regional Anesthesia; Ultrasound
  Arms: Axillary
Procedure: Infraclavicular brachial plexus block — Blocks will be performed under high-resolution real-time ultrasound guidance.
  Patients will be in the supine position. The linear transducer will be initially positioned between the middle and lateral third of the clavicle, scanning on a parasagittal plane.
  The axillary artery and veins will then be sought for. We will try to visualize the three cords of the brachial plexus separately, and to inject local anesthetic around each of them. If this is not possible, the needle will be positioned cranially and posteriorly to the artery, and the injection will be made from there. A 20 G, 17°-bevel needle will be used for all blocks.
  Other Names: Regional Anesthesia; Peripheral nerve block; Ultrasound
  Arms: Infraclavicular

SUMMARY:
This study aims to detect differences in onset time of brachial plexus (i.e., arm) anesthesia using two different nerve block techniques.

Using ultrasound guidance, axillary (i.e., at the armpit) and infraclavicular (i.e., below the collarbone) blocks will be performed to patients undergoing upper limb surgery.

The investigators will analyze how long it takes for anesthesia to be adequate for pain-free surgery, thus determine the optimal technique for this kind of surgery.

DETAILED DESCRIPTION:
Real-time ultrasound guidance has substantially reduced the risk of pneumothorax and/or vascular puncture during infraclavicular brachial plexus blocks. The role of this technique has thus been expanded to overlap those procedures for which an axillary nerve block would be commonly considered as first choice.

A reference block for upper limb surgery thanks to its safety profile and clinical efficacy, the axillary approach may be more painful or unpleasant for some patients.

The investigators aim to determine possible differences in onset time and patient acceptance between the two techniques.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status Class <4
* Scheduled upper extremity orthopedic surgery

Exclusion Criteria:

* Psychiatric or cognitive disorder
* Allergy to study drugs
* Contraindication to nerve block at the assigned site

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-06 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Onset time of brachial plexus sensory block | q5min up to 30 min after the block

SECONDARY OUTCOMES:
Onset of brachial plexus motor block | q5min up to 30 min after the block
Patient satisfaction (3-point scale) | End of surgery
Anesthesia-related procedural pain (0-10 numerical rating scale) | End of block placement
Rescue analgesic requirements during surgery | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Guido Fanelli, MD, Study Chair — Section of Anesthesiology and Critical Care, Dept. of Surgical Sciences, University of Parma; Giorgio Danelli, MD, Principal Investigator — UO II Anestesia e Rianimazione, Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- University Hospital / Azienda Ospedaliero-Universitaria, Parma, PR, Italy